CLINICAL TRIAL: NCT04485494
Title: A Blood Biomarker Study With Clinical Correlation for the Diagnosis and Prognosis of Sports Related Concussion in Elite Rugby
Brief Title: Blood-based Biomarkers for the Prognosis of Sports Related Concussion
Status: Completed | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: CRSU-016
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Traumatic Brain Injury; Sports Injury; Concussion, Mild
Keywords: blood-based biomarker; prognosis; SCAT5; head injury assessment; return to play protocol; sports related concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Athletic Injuries; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples at each time point are taken. Approximately, 30 mL of blood are drawn across 3 vials to allow for collection of whole blood, serum and plasma from the same participant at each time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professional Rugby Athletes: These are the cohort of players that consent to the study and have a preseason baseline blood sample taken. If the participant from this cohort then receives a concussion they are assessed by the World Rugby's Head Injury Assessment (HIA) and then enter into the return to play (RTP) protocol which means they cannot play a competitive game for 6 days.
  Interventions: Diagnostic Test: Biochemical Analysis of Blood Biomarkers

INTERVENTIONS:
Diagnostic Test: Biochemical Analysis of Blood Biomarkers — Using established biochemical techniques, the bloods will be probed for specific biomarkers s100B, UCH-L1, GFAP, and BDNF. The techniques include individual ELISA kits for each biomarker mentioned and Luminex multiplate assay which will probe for all biomarkers in one plate. Ultimately, these techniques will be able to measure the level of these biomarkers in the blood relative to the participants baseline reading.

SUMMARY:
The diagnosis of sports related concussion still relies heavily on a subjective assessment. In this study the investigators want to assess the prognostic value of blood-based biomarkers with recovery from concussive episodes over specific time points post-injury. Our research aims to (1) assess that the World Rugby's head injury assessment (HIA) can identify that a concussion has taken place by measuring specific biomarkers in the blood and (2) to track these biomarkers over time post-injury as a means to assess player health.

DETAILED DESCRIPTION:
The diagnosis and prognosis of sports related concussion (SRC) still rely on a subjective assessment based on the SCAT5 procedure. Our knowledge of how sports related concussion effects an athlete over time is limited as all patients may have different recovery times from concussion. Our research aims to quantitatively confirm that the head injury assessment has predicted a concussion against clinical assessment (SCAT5) and that a return to play protocol allows sufficient recovery time for an athlete.

Numerous novel areas of diagnosis are currently under investigation including protein-based biomarkers. In the context of SRC, these protein biomarkers typically consist of neurological proteins normally confined to the central nervous system or associated with neurological cell damage. Recent studies have compared biomarker levels at different time points post-diagnosis or investigated the relationship between early biomarker levels and return to play (RTP) times. However, the use of these biomarkers for actively evaluating player recovery following SRC has yet to be fully investigated. In this study, the investigators will measure biomarkers levels across multiple time points post-SRC to assess the value of these biomarkers to monitor player recovery. This is of significant for minimising premature RTP and, ultimately, aiming to reduce the chronic long-term effects associated with SRC.

To truly identify a biomarker specific to concussion this study will need to, first, analyse the bloods of concussion patients and compare to the clinical assessment of the head injury assessment (HIA), and, second, measure their levels over time to indicate recovery that may aid in a safe return to play.

Briefly, blood samples are taken from consented participants at the start of pre-season to act as a baseline. Once one of these participants enters the HIA process their bloods are taken post-injury, 6 days after injury and 13 days after injury. Next, the biomarkers are measured in the blood samples at each time point to examine if there is any increase/decrease in their levels.

Study Design:

A prospective cohort study with an uninjured and exercise free control groups.

Population:

All participants are professional rugby players from one professional rugby club were initially invited to participate. Initial contact was made to the Irish Rugby Football Union (IRFU) chief medical officer for permission to run the study over a three-year period. Next permission to run this cohort study was sought from the head coach and medical staff of the professional rugby team.

Baseline Questionnaire:

Participants will complete a baseline questionnaire that includes questions regarding their concussion history including symptoms associated with, length of, and outcome of previous injuries. The questionnaire was developed in line with previous sports-based concussion studies used for ice hockey and Australian football

Timeframes

As part of this study, any participant that enters the standard HIA process will undergo a HIA, a neuropsychometric assessment, and blood sampling at the following time points:

1. Within 72 hours of injury,
2. 6 days post-injury (± 1 day); this aligns with the minimum graduated return to play (GRTP) protocol for a professional rugby player, no player will return to play before 6 days,
3. 13 days post-injury (± 1 day) to examine if biomarkers are still present despite the results the HIA and the neuropsychometric assessment.

Serial HIA Participants that suffer a suspected SRC will complete the HIA protocol at the time points outlined above. This is a form of the SCAT5 which has been modified for professional rugby and GRTP. This assessment will be carried out by the medical officer of the professional rugby club.

Neuropsychometric Assessment During preseason players complete a baseline computed based neuropsychometric assessment - ImPACT. This assessment measures different cognitive domains including visual memory, visual processing speed, reaction times and working memory as well as attention. Post injury players are re-assessed once symptom free to determine recovery fo these domains and to assess for any persistent patterns of deficit. This assessment forms a part of the overall concussion assessment and management plan.

Blood Draw:

The medical officer and/or clinical nurse will take the samples of blood at the timepoints outlined above. The medical officer or nurse usually takes the blood sample from the antecubital vein in the arm.

Bloods are collected by a member of the study team from the medical officer or nurse after the participant has left to ensure confidentiality. Three types of sample vials are used to ensure different types of biochemical techniques can be used and certain markers can be examined; serum, plasma and whole blood. Whole blood samples are immediately aliquoted in 2 mL cryo-vials of 1- 1.5 mL each. For serum samples the blood is allowed to clot within the tube for up to 30 minutes. For both serum and plasma vials, they are centrifuged at 2,000 xg for 10 minutes at 4 °C. The serum and plasma are carefully pipetted and aliquoted into respective 2 mL cryo-vials with no less than 400 µL in each cryo-vial. All aliquoted cryo-vials are placed into storage boxes within a -80 °C freezer for long-term storage. Each aliquot can be removed to probe for different biomarkers without multiple freeze-thaw cycles on the core sample.

Blood Biomarkers The blood-based biomarkers that can be analysed using standard biochemical techniques for a targeted and hypothesis-based procedures using ELISA kits or Luminex multiplex assays. Serum and plasma samples allows for a multitude of targets to be analysed which may be found in either serum or plasma. For this type of analysis common targets can be used to compare across the timepoints. The biomarkers under investigation can be but not limited to s100β, ubiquitin carboxyl-terminal hydrolase isoenzyme L1, glial fibrillar acidic protein and total, Tau protein and Brain-derived neurotrophic factor.

Outcomes Each participant that is believed to have a SRC will enter the HIA process. These participants will have clinical assessments conducted at pre-defined time points, in line with the World Rugby guidelines. Blood samples will also be acquired at these time points to quantify the levels of blood-based biomarkers. Biomarker levels will be correlated to the results of the HIA and neuropsychometric assessments. This will facilitate preliminary investigation of the correlation between clinical assessments and biomarker levels to determine if the biomarkers can be used to objectively assess SRC recovery

Investigations:

A collaborative relationship exists between this research group and the University of Limericks (UL) Clinical Research Support Unit (CRSU). The CRSU provided advice and supported the delivery of this research project to the highest standard of research and clinical governance in accordance with the requirements of ICH Good Clinical Practice (ICH-GCP) Guidelines and all applicable regulatory requirements. The participant contact element of this study was conducted by adhering to the CRSU's Quality Management System (QMS).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to participate if they

1. are part of the professional rugby team's senior squad or the academy;
2. aged over 18;
3. consent to the study over the whole season.

Exclusion Criteria:

Participants are excluded if they

1. are unable to attend the preseason baseline draw;
2. unable to give informed consent.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants are professional rugby players from a professional rugby club were have been invited to participate. Initial contact was made to the Irish Rugby Football Union (IRFU) chief medical officer for permission to run the study over a three-year period. Next permission to run this cohort study was sought from the head coach and medical staff of the professional rugby team.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical Diagnosis | Bloods to be taken within 72 hours of injury
  Measure the levels of blood biomarkers in rugby players that have experienced a concussion, confirmed via HIA and neuropsychometric assessment, to assess the utility of these biomarkers for concussion diagnosis
Clinical Recovery | Bloods to be taken within 6 and 13 days post-injury
  Track the levels of the blood biomarkers over time, post-injury to determine if biomarker levels correlate with clinical recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Kearns, MD, Principal Investigator — Munster Rugby
Locations (1):
- Munster Rugby, Limerick, Munster, Ireland

REFERENCES:
- [Background] Fuller CW, Taylor A, Kemp SP, Raftery M. Rugby World Cup 2015: World Rugby injury surveillance study. Br J Sports Med. 2017 Jan;51(1):51-57. doi: 10.1136/bjsports-2016-096275. Epub 2016 Jul 26. PMID 27461882
- [Background] McCrea M, Meier T, Huber D, Ptito A, Bigler E, Debert CT, Manley G, Menon D, Chen JK, Wall R, Schneider KJ, McAllister T. Role of advanced neuroimaging, fluid biomarkers and genetic testing in the assessment of sport-related concussion: a systematic review. Br J Sports Med. 2017 Jun;51(12):919-929. doi: 10.1136/bjsports-2016-097447. Epub 2017 Apr 28. PMID 28455364
- [Background] Papa L. Potential Blood-based Biomarkers for Concussion. Sports Med Arthrosc Rev. 2016 Sep;24(3):108-15. doi: 10.1097/JSA.0000000000000117. PMID 27482776
- [Background] O'Connell B, Kelly AM, Mockler D, Oresic M, Denvir K, Farrell G, Janigro D, Wilson F. Use of Blood Biomarkers in the Assessment of Sports-Related Concussion-A Systematic Review in the Context of Their Biological Significance. Clin J Sport Med. 2018 Nov;28(6):561-571. doi: 10.1097/JSM.0000000000000478. PMID 29035978
- [Background] Jeter CB, Hergenroeder GW, Hylin MJ, Redell JB, Moore AN, Dash PK. Biomarkers for the diagnosis and prognosis of mild traumatic brain injury/concussion. J Neurotrauma. 2013 Apr 15;30(8):657-70. doi: 10.1089/neu.2012.2439. PMID 23062081
- [Background] Di Battista AP, Rhind SG, Baker AJ, Jetly R, Debad JD, Richards D, Hutchison MG. An investigation of neuroinjury biomarkers after sport-related concussion: from the subacute phase to clinical recovery. Brain Inj. 2018;32(5):575-582. doi: 10.1080/02699052.2018.1432892. Epub 2018 Feb 8. PMID 29420083
- [Background] Shahim P, Tegner Y, Marklund N, Blennow K, Zetterberg H. Neurofilament light and tau as blood biomarkers for sports-related concussion. Neurology. 2018 May 15;90(20):e1780-e1788. doi: 10.1212/WNL.0000000000005518. Epub 2018 Apr 13. PMID 29653990
- [Background] Ercole A, Thelin EP, Holst A, Bellander BM, Nelson DW. Kinetic modelling of serum S100b after traumatic brain injury. BMC Neurol. 2016 Jun 17;16:93. doi: 10.1186/s12883-016-0614-3. PMID 27315805
- [Derived] Kearns J, Ross AM, Walsh DR, Cahalane RM, Hinchion R, Ryan MC, Conway E, Comyns TM, Kenny IC, O'Connor EM, McGourty KD, Mulvihill JJE. A blood biomarker and clinical correlation cohort study protocol to diagnose sports-related concussion and monitor recovery in elite rugby. BMJ Open Sport Exerc Med. 2020 Nov 26;6(1):e000948. doi: 10.1136/bmjsem-2020-000948. eCollection 2020. PMID 34422289

DOCUMENTS (1):
  • Informed Consent Form (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04485494/ICF_000.pdf